CLINICAL TRIAL: NCT03645668
Title: Efficacy and Pharmacokinetics of Meropenem in Different Administration for Patients With Severe Sepsis
Brief Title: Efficacy and Pharmacokinetics of Meropenem in Severe Septic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-18-003
Record Dates: First submitted 2018-02-07; First posted 2018-08-24 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Sepsis
Keywords: sepsis，meropenem，2 steps administration
MeSH Terms: conditions — Sepsis | interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): meropenem injection, 1.0g, q8h,intravenous infusion ,0.5g/0.5h+0.5g/4h
  Interventions: Drug: Meropenem Injection
- Control group (Other): meropenem injection, 1.0g, q8h,continuous intravenous infusion duration ,1h
  Interventions: Drug: Meropenem Injection

INTERVENTIONS:
Drug: Meropenem Injection — Different administration types between two groups
  Other Names: meropenem,MEPEM

SUMMARY:
The experimental and control group were used different administration of Meropenem through monitoring the Meropenem plasma concentration and clinical data

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial, which the subjects were severe sepstic patients for selecting Meropenem as antimicrobial drugs. The experimental and control group were used different administration of Meropenem through monitoring the Meropenem plasma concentration and clinical data, eventually demonstrate the effecacy and safety of Meropenem in patients with severe infection and optimize the best clinical practice for antimicrobial agents.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients, whose informed consent has been obtained;
2. Clinical diagnosis of Sepsis

Exclusion Criteria:

1. Pregnancy or lactation;
2. Treated with other carbapenems;
3. Cannot be evaluated for efficacy and safety result from lack of clinical and laboratory parameter for Infection assessment;
4. Allergy to meropenem or other β-lactams, or the history of allergy;
5. Resistant to meropenem according to the antimicrobial susceptibility test;
6. Epilepsy or history of epilepsy;
7. History of seizures;
8. Combined medicine with sodium valproate;
9. Combined medicine with anti-MRSA, anti-fungal drugs;
10. with severe liver or renal dysfunction;
11. Terminal cancer;
12. Septic shock;
13. APACH II ≥20;
14. Inappropriate to participate in the trial evaluated by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
T>MIC | Day 1
  Time above MIC% per administration interval

SECONDARY OUTCOMES:
APACHE II score | Day 0,Day 4,Day 8
  Change of Acute physiology and chronic health evaluation score (APACHE II score) during period of treatment
SOFA | Day 0,Day 4,Day 8
  Change of Sepsis-related Organ Failure Assessment score (sofa) during period of treatment
Mortality | Day 28
  Mortality within 28 days
highest temperature | Day 0,Day 4,Day 8
  Variation of the highest temperature

CONTACTS AND LOCATIONS:
Overall Officials: Aihua FEI, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality, China